CLINICAL TRIAL: NCT00428493
Title: Prospective Study of Individuals Exposed to Confirmed Cases of Human Influenza A (H5N1) Infection in China
Brief Title: Prospective Study of AI H5N1 in China
Status: Completed | Type: Observational
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Other Study IDs: 06-0055
Record Dates: First submitted 2007-01-25; First posted 2007-01-30 (Estimated); Last update posted 2008-05-30 (Estimated); Status verified 2008-05

CONDITIONS: Influenza
Keywords: human influenza A, H5N1, bird flu, avian influenza, China
MeSH Terms: conditions — Influenza, Human; Influenza in Birds

STUDY DESIGN:
Time Perspective: Prospective

SUMMARY:
The purpose of this study is to see if people in China who have contact with someone infected with bird flu (H5N1) become infected themselves without necessarily getting sick. Adults and children greater than 1 year of age who have contact with someone infected with bird flu may participate in the study. At the first 1-2 study visits, a blood sample will be taken from volunteers in order to test for antibodies, the part of the blood that fights infection. If the result of the H5N1 antibody test is positive after the 1st or 2nd study visit, an additional blood sample will be collected during a 3rd and 4th study visit. Volunteers will be asked questions about their work, home life, and possible contact with poultry, other birds, animals, and people infected with bird flu. Participants will be involved in study related procedures for up to 90 days.

DETAILED DESCRIPTION:
This will be a prospective cohort study of individuals exposed to confirmed cases of Human Influenza A (H5N1) infection in China. The study will be conducted over a period of approximately one year. Adults and children, greater than age 1, who meet the eligibility criteria will be consented and enrolled in the study. These subjects will undergo up to two blood draws for serologic testing of the presence of H5N1 antibodies according to an algorithm. These subjects will also be administered a structured questionnaire for collection of demographic information, information on potential exposure to poultry, other birds or animals, or infected humans and any clinical symptoms. This questionnaire will have similar data elements to the questionnaires used in the past for collection by the China CDC. The questionnaires were administered in areas of China where there have been poultry and human cases, as well as, other high risk populations in non-outbreak areas. Enrolled participants will complete two study visits no more than one month apart with a third visit for those who test positive for influenza A H5N1 infection. Participants who consent to HIV testing will have a fourth visit to obtain their HIV test results. The primary study objective is to determine the prevalence of antibodies to avian influenza A (H5N1) virus among close contacts and health care workers associated with confirmed H5N1 infected individuals in China. The secondary study objectives are to: describe risk factors for human infection with avian influenza A (H5N1) virus in China; evaluate the incidence of seroconversion and increases in titer of H5N1 antibodies; describe risk factors associated with seroconversion and increases in titer of H5N1 antibodies; determine T-cell immune responses in H5N1 infected individuals; and determine the prevalence of co-infection of H5N1 and HIV-1. The primary endpoint is detection of avian influenza H5N1 infection as determined by a positive result on Hemagglutination Inhibition (HI) and confirmed by Microneutralization (MN). Corresponding with the secondary study objectives, the following will be assessed as secondary study endpoints: association of risk factors with avian influenza seropositivity, including demographic characteristics and various exposures to poultry, other birds, and to infected humans; H5N1 serum antibody titer seroconversion or a greater than or equal to 4-fold increase in titer; association of risk factors with avian influenza seroconversion, including demographic characteristics and various exposures to poultry, other birds, and to infected humans; HIV-1 infection as determined by ELISA and Western Blot assays and co-infection of H5N1 and HIV-1 as determined by both assays described above; and T-cell responses to H5N1 as determined by ELISPOT assay and ICS.

ELIGIBILITY:
Inclusion Criteria:

1. Informed consent for study participation provided by the volunteer or, for children, by a parent or legal guardian. Children aged 10-18 will be asked to assent.
2. Adults and children > 1 year old.
3. Close contacts or health care worker of confirmed human H5N1 case.

Exclusion Criteria:

1. Children under 12 months old.

Min Age: 12 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 4000
Dates: Start 2007-01; Study Completion 2008-01

CONTACTS AND LOCATIONS:
Locations (1):
- Chinese Center for Disease Control and Prevention, Beijing, China